CLINICAL TRIAL: NCT05750472
Title: Neck Awareness, Cognitive Function and Left/Right Judgment Performance in Individuals With Neck Pain: A Cross-sectional Study
Brief Title: Left/Right Neck Judgment Performance in Individuals With Neck Pain
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Aysegul Bostan, Research Assistant, Bahçeşehir University
Other Study IDs: BAU-AYSEGULBOSTAN-002
Record Dates: First submitted 2023-01-30; First posted 2023-03-01 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain
Keywords: Proprioception; Cognitive Function; Neck Pain; Body Images; Imagery
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neck Pain Group: group evaluated with scales
- Healthy Group: group evaluated with scales

SUMMARY:
Neck pain is one of the leading causes of disability worldwide and ranks fourth among the pathologies that result in disability. Although neck pain can be attributed to traumatic or inflammatory disorders, the majority of neck pain has no discernible cause and is considered idiopathic. Neck pain that lasts longer than 3 months takes the form of chronic neck pain. Some problems such as changes in muscle behavior and decrease in proprioceptive sensory input are observed in individuals with chronic neck pain. The presence of such problems, especially the dysfunction of the deep cervical muscles and the inability of the proprioceptors to provide motor control, cause the position sense to be impaired in these individuals and the awareness of the neck of the individuals decreases.

The Left Right Judgment Task (LRJT) is a form of implicit motor imagery that involves determining as accurately and quickly as possible whether an image of a body part belongs to the left or right side. LRJT performance differences have been hypothesized to reflect changes in central nervous system functioning, errors in judgment, and changes in bodily representations. It has been shown that LRJT is a complex mental task that includes cognitive, sensory, motor and behavioral processes and can be associated with them.

Recent studies have revealed that neck pain causes proprioceptive disorder and that proprioceptive training should be done in these individuals. A study showed that there is a strong correlation between biasedness judgment accuracy and proprioception.

In this context, the investigators aimed to investigate the knowledge about the effect of individuals with neck pain on proprioception, cortical body diagram and pain.

DETAILED DESCRIPTION:
Method:

The demographic characteristics of individuals who come to the clinic with a complaint of neck pain and meet the inclusion criteria as directed by the doctor will be recorded. The level of neck involvement will be determined according to the Neck Paint Task Force. Functionality level of all participants will be evaluated by Neck Disability Index, pain intensity by Visual Analog Scale, fear of movement by Tampa Kinesiophobia Scale, body awareness by left/right neck rotation, judgment task performance and neck awareness by Fremantle Neck Awareness Questionnaire.

Left/right neck rotation decision task performance With the Recognise™ (http://www.nongroup.com/Recognise) application, the participant will be asked to do it on a single type tablet provided by the physiotherapist. After participants practice on 10 images before proceeding to the main tasks, 40 images will be displayed on the tablet screen in random order at five-second intervals. The participant will decide and answer as soon as possible whether the picture is right or left. The average percentage and reaction time of correctly identified images on both sides will then be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who do not experience neck or back pain that interferes with their normal activities, or pain responsible for disability.
* No previous medical intervention or treatment for a neck problem.

Exclusion Criteria:

* To have received treatment in the last 6 months
* He had neck surgery
* Suspicion of malignant or systemic disease
* Neurological disease or injury
* Vertigo, nausea, visual disturbances,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with neck pain and healthy controls
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The Left Right Neck Judgment Task | First day
  RecogniseTM Hands is an app designed for both iPhone and iPad. As part of a graded motor imagery rehabilitation program, left/right hand discrimination measures decision-making accuracy.
  The Recognise™ (NOI, Adelaide, Australia) application used in individuals with neck pain to examine the applicability of left /right neck discrimination decision making in neck patients, and it was found to be appropriate. In this context, data will be collected through the Recognise™ (NOI, Adelaide, Australia) application in this study. Individuals will look at the pictures displayed on the online computer and respond to each picture by stating whether the head of the model in the picture is facing left or right relative to their shoulders. Participants are asked to respond as quickly as possible without guessing.
Pain Intensity | First day
  Pain intensity of individuals will be evaluated subjectively with Visual Analog Scale. This scale consists of a 10 cm linear line. The starting point of the line is 0, no pain; endpoint of 10, the most severe pain encountered in life; 5 indicates moderate pain. Individuals will be asked to rate the severity of their pain numerically on the scale.

SECONDARY OUTCOMES:
Kinesiophobia | First day
  Fear of movement will be evaluated with the Tampa kinesiophobia scale. Tampa kinesiophobia scale is a 17-item questionnaire developed by Koretal in 1991 for musculoskeletal pain. This scale includes the parameters of injury/re-injury and fear avoidance in related activities. Each question on this scale was scored as (1 = disagree, 4 = strongly agree). While scoring, items 4, 8, 12 and 16 are reversed and then the total score is obtained. The person gets a total score between 17-68.

OTHER OUTCOMES:
Evaluation of Neck Disability | First day
  The effect of chronic neck pain on activities of daily living was evaluated with the Neck Disability Index. The index, which evaluates subjective symptoms and activities of daily living, consists of 10 sections (pain severity, personal care, lifting, reading, headache, concentration, work life, driving, sleep and leisure activities). There are 6 options for each section, ranging from 0 to 5 points. The total score ranges from 0 to 50 (0: no disability; 50: maximum disability), and an increase in the total score indicates an increase in disability. In the evaluation of our study, the percentage of each score was calculated by taking the percentage of each score in order to obtain an equal score distribution in case the patients did not answer some questions. 8 percent and six "no apologies" were accepted.

CONTACTS AND LOCATIONS:
Overall Officials: Rsch Asst Aysegul Bostan, PhD candid, Principal Investigator — Bahçeşehir University; PT Bedia Ozdemir, MSc Candid, Principal Investigator — Arel University; Prof. Ozlem Ulger, Professor, Study Director — Hacettepe University
Locations (1):
- Bahcesehir Universty, Istanbul, Besiktas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Popescu A, Lee H. Neck Pain and Lower Back Pain. Med Clin North Am. 2020 Mar;104(2):279-292. doi: 10.1016/j.mcna.2019.11.003. Epub 2019 Dec 20. PMID 32035569
- [Background] Stanton TR, Leake HB, Chalmers KJ, Moseley GL. Evidence of Impaired Proprioception in Chronic, Idiopathic Neck Pain: Systematic Review and Meta-Analysis. Phys Ther. 2016 Jun;96(6):876-87. doi: 10.2522/ptj.20150241. Epub 2015 Oct 15. PMID 26472296
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Falla D, Bilenkij G, Jull G. Patients with chronic neck pain demonstrate altered patterns of muscle activation during performance of a functional upper limb task. Spine (Phila Pa 1976). 2004 Jul 1;29(13):1436-40. doi: 10.1097/01.brs.0000128759.02487.bf. PMID 15223935
- [Background] Curtis BR, Fitchett E. A vascular cause of neck pain. Intern Emerg Med. 2017 Sep;12(6):895-897. doi: 10.1007/s11739-016-1592-6. Epub 2016 Dec 24. No abstract available. PMID 28013445
- [Background] Malmstrom EM, Westergren H, Fransson PA, Karlberg M, Magnusson M. Experimentally induced deep cervical muscle pain distorts head on trunk orientation. Eur J Appl Physiol. 2013 Oct;113(10):2487-99. doi: 10.1007/s00421-013-2683-y. Epub 2013 Jun 29. PMID 23812089
- [Background] Alahmari KA, Reddy RS, Silvian P, Ahmad I, Nagaraj V, Mahtab M. Influence of chronic neck pain on cervical joint position error (JPE): Comparison between young and elderly subjects. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1265-1271. doi: 10.3233/BMR-169630. PMID 28800305
- [Background] Osuagwu BA, Vuckovic A. Similarities between explicit and implicit motor imagery in mental rotation of hands: an EEG study. Neuropsychologia. 2014 Dec;65:197-210. doi: 10.1016/j.neuropsychologia.2014.10.029. Epub 2014 Oct 30. PMID 25446966
- [Background] 10. Moseley G. L. The Graded Motor Imagery Handbook. Noigroup publications; 2012.
- [Background] Pelletier R, Bourbonnais D, Higgins J, Mireault M, Danino MA, Harris PG. Left Right Judgement Task and Sensory, Motor, and Cognitive Assessment in Participants with Wrist/Hand Pain. Rehabil Res Pract. 2018 Aug 26;2018:1530245. doi: 10.1155/2018/1530245. eCollection 2018. PMID 30225144
- [Background] Peng B, Yang L, Li Y, Liu T, Liu Y. Cervical Proprioception Impairment in Neck Pain-Pathophysiology, Clinical Evaluation, and Management: A Narrative Review. Pain Ther. 2021 Jun;10(1):143-164. doi: 10.1007/s40122-020-00230-z. Epub 2021 Jan 12. PMID 33464539
- [Background] Elsig S, Luomajoki H, Sattelmayer M, Taeymans J, Tal-Akabi A, Hilfiker R. Sensorimotor tests, such as movement control and laterality judgment accuracy, in persons with recurrent neck pain and controls. A case-control study. Man Ther. 2014 Dec;19(6):555-61. doi: 10.1016/j.math.2014.05.014. Epub 2014 Jun 10. PMID 24957711
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] Davidson CJ, Ganion LR, Gehlsen GM, Verhoestra B, Roepke JE, Sevier TL. Rat tendon morphologic and functional changes resulting from soft tissue mobilization. Med Sci Sports Exerc. 1997 Mar;29(3):313-9. doi: 10.1097/00005768-199703000-00005. PMID 9139169
- [Background] Telci EA, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagli N. The cultural adaptation, reliability, and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2009 Jul 15;34(16):1732-5. doi: 10.1097/BRS.0b013e3181ac9055. PMID 19770615
- [Background] Wand BM, Catley MJ, Rabey MI, O'Sullivan PB, O'Connell NE, Smith AJ. Disrupted Self-Perception in People With Chronic Low Back Pain. Further Evaluation of the Fremantle Back Awareness Questionnaire. J Pain. 2016 Sep;17(9):1001-12. doi: 10.1016/j.jpain.2016.06.003. Epub 2016 Jun 18. PMID 27327235
- [Background] Onan D, Gokmen D, Ulger O. The Fremantle Neck Awareness Questionnaire in Chronic Neck Pain Patients: Turkish Version, Validity and Reliability Study. Spine (Phila Pa 1976). 2020 Feb 1;45(3):E163-E169. doi: 10.1097/BRS.0000000000003207. PMID 31425430
- [Background] Haldeman S, Carroll L, Cassidy JD, Schubert J, Nygren A; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. The Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders: executive summary. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S5-7. doi: 10.1097/BRS.0b013e3181643f40. No abstract available. PMID 18204400
- [Background] 20. Yılmaz Ö.T, Yakut Y, Uygur F, Uluğ N. Tampa kinezyofobi ölçeği"nin Türkçe versiyonu ve test-tekrar test güvenirliği. Fizyoterapi Rehabilitasyon 2011;22(1):44-49.
- [Background] Moseley GL. Why do people with complex regional pain syndrome take longer to recognize their affected hand? Neurology. 2004 Jun 22;62(12):2182-6. doi: 10.1212/01.wnl.0000130156.05828.43. PMID 15210879
- [Background] Wallwork SB, Butler DS, Fulton I, Stewart H, Darmawan I, Moseley GL. Left/right neck rotation judgments are affected by age, gender, handedness and image rotation. Man Ther. 2013 Jun;18(3):225-30. doi: 10.1016/j.math.2012.10.006. Epub 2013 Jan 26. PMID 23357411